CLINICAL TRIAL: NCT00754585
Title: The Effectiveness of the Logic Back™Support in Promoting a Comfortable Neutral Low Back Position, Reduced Muscular Effort, Improved Performance, and Decreased Postural Shifts in Seating.
Brief Title: The Effectiveness of the Logic Back™Support.
Status: Completed | Type: Observational
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: Logic Back (Unknown); McMaster University (Other)
Responsible Party: John J. Triano, DC, PhD, Canadian Memorial Chiropractic College
Other Study IDs: 082007
Record Dates: First submitted 2008-09-04; First posted 2008-09-18 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Low Back Pain; Posture
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I: All participants will perform the five Chair Support tasks: (1) quiet standing, sitting, (2) upper back unsupported, (3) sitting, upper back unsupported with Logic Back in place, (4) sitting in a standard ergonomic chair, and (5) sitting in a standard ergonomic chair with Logic Back in place. Aside from the Quiet Standing trials which will be performed first, the order of Chair Support will be randomized. Participants will perform the Chair Support task for 30 minutes while quietly watching a movie DVD of their choice. The DVDs provided will the "light" in content without a lot of suspense or emotion. Data will be collected for the final two minutes of each 30-minute trial.
  Interventions: Device: Logic Back Grahl Duo Back Model DB11-01

INTERVENTIONS:
Device: Logic Back Grahl Duo Back Model DB11-01 — The device is placed against the back rest of a chair. The tension of the straps are adjusted for each participant to obtain the ENP.

SUMMARY:
Back pain and chair use are the second most important health factors for the aging workforce. Besides personal suffering, postural discomfort in the workplace reduces performance and productivity, both of which can be improved by raising comfort levels. In an attempt to improve comfort and reduce injury risk, ergonomic chairs are commonly equipped with lumbar supports in an attempt to support a "neutral" spine. However, people often alter their position when such a device is in place as they arch their back to conform to it. The Logic Back support offers a simple means to alter posture and reduce associated strain on the lower back during seated tasks by supporting the "Effortless Neutral Position" or the natural curvature of the low back. Although it has been used clinically by many practitioners, its effectiveness has yet to be shown by scientific study. The current work will help to understand if and why the Logic Back is effective and how it can become a low-cost solution to reduce the discomfort of those suffering from low back pain.

The purpose of this study is to determine the effectiveness of the Logic Back and the "Effortless Neutral Position" in improving comfort and functional performance during seated tasks, as compared to a standard, ergonomic chair.

DETAILED DESCRIPTION:
Seventeen of the top Canadian occupations typically have workers sitting a significant proportion of their work day. An average of 30% of Ontario WSIB lost time claims since 1996 involve low back injury. The return to work objective for twenty percent of these patients requires prolonged sitting in their work stations. While a number of these studies have claimed a relationship between sitting and LBP, the relationship is complex. Back pain and chair use are the second most important health factors for the aging workforce. The odds ratio for LBP is estimated for seated tasks at 1.9721. Prolonged and monotonous, low-level mechanical loads associated with a seated posture are thought to provoke pain.

Besides personal suffering, postural discomfort in the workplace reduces performance and productivity, both of which can be improved by raising comfort levels. According to Corlett (2006), other lumbar supports do not exert enough pressure on the spine to actually change its configuration. However, the patient often alters their posture when such a device is in place as they arch their back to conform to it. The Logic Back support offers a simple means to alter posture and reduce associated strain on the lower back during seated tasks by promoting the neutral standing lordotic posture. Clinically, it has been shown to support the ENP or the natural standing lordotic posture. Although its clinical applicability has been accepted by many practitioners, its effectiveness in improving seated comfort and functional task performance has yet to be quantified in LBP patients who perform seated tasks. This study will help to understand why the Logic Back or ENP must be considered when planning return-to-work goals and methods to reduce first-time injury incidence in the workplace.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between ages of 20-55
* With or without lower back pain

Exclusion Criteria:

* Participants currently experiencing neck, shoulder or arm pain
* Participants who have low back pain of non-musculoskeletal origin

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Males only, ages between 20-55 years of age
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Seated CoP Shift Rate: The CoP wil be measured by use of a TEKSCAN CONFORMat system - a thin sensing mat that is placed on the chair surface and measures the relative pressure applied by the legs and buttocks during seated tasks. | 30 minutes
Functional Performance (Task Repetition Frequency)- three dynamic, seated performance tests are used and include: Test 1 - "Waist level-Up", Test 2 - "Eye level-down", and Test 3 - "Overhead work". | 5 minutes

SECONDARY OUTCOMES:
Self-Reports of Comfort: Tests such as the Visual Analog Scale (VAS) or mapping by body area will be used. Participants will also be asked to record their current level of discomfort on a 10cm VAS for each body area. | 5 minutes
Postural Quantification: Electromagnetic sensors (Polhemus 3-space Isotrak system) will allow for the continuous and automatic monitoring of key body landmark positions and orientations in space. | 2 minutes
RMS-EMG (Muscular Exertion): Following standard skin preparation (shaving as needed, alcohol cleansing and mild abrasion) surface electrodes (10 mm Ag-AgCL, 1 cm interspace) will be applied and oriented parallel to the target muscles. | 2 minutes
Evaluation of Spinal Loads: Load on the spine is a combined effect of the posture, muscle activity and task being performed. The UM3D model is a validated lift task analysis system. | 2 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Canadian Memorial Chiropractic College, North York, Ontario

REFERENCES:
- [Derived] Grondin DE, Triano JJ, Tran S, Soave D. The effect of a lumbar support pillow on lumbar posture and comfort during a prolonged seated task. Chiropr Man Therap. 2013 Jul 4;21(1):21. doi: 10.1186/2045-709X-21-21. PMID 23826832